CLINICAL TRIAL: NCT06299163
Title: A Phase 1 Study of NM32-2668 (Anti-ROR1/CD3/Anti-HSA Tri-Specific Antibody) in Adult Patients With Selected Advanced Solid Tumors
Brief Title: NM32-2668 in Adult Patients With Selected Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision
Sponsor: Numab Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NB-NM032-2668-101
Record Dates: First submitted 2024-02-26; First posted 2024-03-07 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Ovarian Carcinoma; Fallopian Tube Carcinoma; Peritoneal Carcinoma; Endometrial Cancer; Adenocarcinoma of Lung; Triple Negative Breast Cancer; Liposarcoma; Leiomyosarcoma; Mesothelioma, Malignant; Adenocarcinoma - Gastroesophageal Junction (GEJ); Adenocarcinoma of the Stomach; Melanoma, Malignant; Renal Cell Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Endometrial Neoplasms; Adenocarcinoma of Lung; Triple Negative Breast Neoplasms; Liposarcoma; Leiomyosarcoma; Mesothelioma, Malignant; Melanoma; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- NM32-2668 (Experimental)
  Interventions: Biological: NM32-2668

INTERVENTIONS:
Biological: NM32-2668 — Anti-ROR1/Anti-Cluster of Differentiation 3 (CD3)/Anti-Human Serum Albumin (HSA) Tri-Specific Antibody

SUMMARY:
This is a first-in-human, open-label, multi-center, Phase 1, dose-escalation study with expansion cohorts to evaluate NM32-2668 for safety and immunogenicity, to determine the maximal tolerated dose and recommended Phase 2 dose, define the pharmacokinetics, to explore the pharmacodynamics, and to obtain preliminary evidence of the clinical activity in adult patients with selected advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed, advanced-stage protocol-specified solid tumors.
* Confirmed ROR1 tumor expression.
* Patients who have undergone at least one prior systemic therapy and have radiologically or clinically determined progressive disease during or after most recent line of therapy, and for whom no further standard therapy is available, or who are intolerable or have medical contraindications to standard therapy.

Exclusion Criteria:

* Prior treatment with any agent targeting ROR1 or prior treatment with a CD3 T-cell engaging therapy.
* Prior treatment with chimeric antigen receptor (CAR) cell therapy within 90 days prior to first dose of NM32-2668.
* Systemic anti-neoplastic therapy within five half-lives or 21 days, whichever is shorter, prior to first dose of NM32-2668.
* Wide-field radiotherapy (> 30% of marrow-bearing bones) within 28 days, or focal radiation for analgesic purpose or for lytic lesions at risk of fracture within 14 days prior to first dose of NM32-2668, or no recovery from side effects of such prior interventions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) | Through 28 days post-infusion
Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) as assessed by CTCAE v5.0 / ASTCT (for Cytokine Release Syndrome [CRS]) | Through 50 days post-final dose administration
Frequency of dose interruptions/reductions | Up to 12 treatment cycles or through treatment discontinuation, whichever occurs first
Duration of dose interruptions/reductions | Up to 12 treatment cycles or through treatment discontinuation, whichever occurs first

SECONDARY OUTCOMES:
Assessment of the maximum observed serum concentration (Cmax) | From date of randomization until end of treatment, assessed for up to 336 days (i.e., 12 treatment cycles) or through treatment discontinuation
Assessment of the the minimum observed serum concentration (Cmin) | From date of randomization until end of treatment, assessed for up to 336 days (i.e., 12 treatment cycles) or through treatment discontinuation
Time from dosing at which maximum observed serum concentration is apparent (Tmax) | From date of randomization until end of treatment, assessed for up to 336 days (i.e., 12 treatment cycles) or through treatment discontinuation
Assessment of the terminal phase (apparent elimination) rate constant (λz) | From date of randomization until end of treatment, assessed for up to 336 days (i.e., 12 treatment cycles) or through treatment discontinuation
Assessment of the elimination half-life (t½) | From date of randomization until end of treatment, assessed for up to 336 days (i.e., 12 treatment cycles) or through treatment discontinuation
Assessment of the area under the serum concentration-time curve extrapolated from the last quantifiable concentration to infinity (AUC[0-infinity]) | From date of randomization until end of treatment, assessed for up to 336 days (i.e., 12 treatment cycles) or through treatment discontinuation
Assessment of the area under serum concentration-time curve over dosing interval (AUCtau) | From date of randomization until end of treatment, assessed for up to 336 days (i.e., 12 treatment cycles) or through treatment discontinuation
Assessment of clearance (CL) of NM32-2668 in serum | From date of randomization until end of treatment, assessed for up to 336 days (i.e., 12 treatment cycles) or through treatment discontinuation
Assessment of the volume of distribution (Vd) of NM32-2668 in serum | From date of randomization until end of treatment, assessed for up to 336 days (i.e., 12 treatment cycles) or through treatment discontinuation
Assessment of accumulation ratios of Cmax (ARcmax) of NM32-2668 in serum | From date of randomization until end of treatment, assessed for up to 336 days (i.e., 12 treatment cycles) or through treatment discontinuation
Assessment of accumulation ratios of Cmin (ARcmin) of NM32-2668 in serum | From date of randomization until end of treatment, assessed for up to 336 days (i.e., 12 treatment cycles) or through treatment discontinuation
Assessment of accumulation ratios of AUC (ARauc) of NM32-2668 in serum | From date of randomization until end of treatment, assessed for up to 336 days (i.e., 12 treatment cycles) or through treatment discontinuation
Frequency of specific anti-drug antibodies (ADAs) to NM32-2668 | From date of randomization until end of treatment, assessed for up to 336 days (i.e., 12 treatment cycles) or through treatment discontinuation
Concentration of specific ADAs to NM32-2668 | From date of randomization until end of treatment, assessed for up to 336 days (i.e., 12 treatment cycles) or through treatment discontinuation
Incidence of specific ADAs by category to NM32-2668 | From date of randomization until end of treatment, assessed for up to 336 days (i.e., 12 treatment cycles) or through treatment discontinuation
Best Overall Response (BOR) according to RECIST 1.1 | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed for up to 30 days following last dose of study treatment
Overall Response Rate (ORR) according to RECIST 1.1 | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed for up to 30 days following last dose of study treatment
Disease Control Rate (DCR) according to RECIST 1.1 | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed for up to 30 days following last dose of study treatment
Progression-free Survival (PFS) according to RECIST 1.1 | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed through study completion (on average, 1 year after last treatment)
Time to Response (TTR) according to RECIST 1.1 | From date of randomization until the date of first documented treatment response according to RECIST 1.1
Duration of Response (DOR) according to RECIST 1.1 | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed through study completion (on average, 1 year after last treatment)
Overall Survival (OS) | From date of randomization until the date of death from any cause, assessed through study completion (on average, 1 year after last treatment)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - The University of Chicago Medical Center (UCMC), Chicago, Illinois
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh Medical Center (UPMC) - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Lifespan Cancer Institute at Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin